CLINICAL TRIAL: NCT06004336
Title: A Randomized Trial of Maintenance Systemic Therapy After Radiation for Oligometastatic Renal Cell Carcinoma (ASTROs)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0006; NCI-2023-06314 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Oligometastatic Renal Cell Carcinoma
MeSH Terms: interventions — pembrolizumab; Radiotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Radiation therapy (Control Arm) (Experimental): Participants will be asked to receive radiation therapy and be randomly assigned to receive pembrolizumab or not after that.
  Interventions: Drug: Pembrolizumab; Radiation: Radiation therapy
- Radiation Therapy and Pembrolizumab (Experimental): Participants will be asked to receive radiation therapy and be randomly assigned to receive pembrolizumab or not after that.
  Interventions: Drug: Pembrolizumab; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Pembrolizumab — Given by vein (IV)
Radiation: Radiation therapy — Given by vein (IV)

SUMMARY:
To learn if adding 1 year of therapy with pembrolizumab can help to continue to control RCC after radiation therapy.

DETAILED DESCRIPTION:
Primary Objectives:

* To evaluate PFS in patients randomized to definitive RT followed by pembrolizumab versus definitive RT followed by observation.

Secondary Objectives:

Secondary Objective #1:

* To evaluate overall survival (OS) in patients randomized to definitive RT followed by maintenance pembrolizumab versus definitive RT followed by observation.

Secondary Objective #2:

* To evaluate time to next line systemic therapy (defined as systemic therapy given after pembrolizumab) in patients randomized to definitive RT followed by maintenance pembrolizumab versus definitive RT followed by observation.

Secondary Objective #3:

* To evaluate local recurrence free survival (LRFS) in patients randomized to definitive RT followed by maintenance pembrolizumab versus definitive RT followed by observation.

Secondary Objective #4:

* To evaluate distant recurrence free survival (DRFS) in patients randomized to definitive RT followed by maintenance pembrolizumab versus definitive RT followed by observation.

Secondary Objective #5:

* To evaluate estimate PFS2, LRFS2, and DRFS2 in patients who crossed over from one randomization arm to the other arm.

Secondary Objective #6:

* To evaluate frequency of adverse events (AEs) in patients randomized to definitive RT followed by maintenance pembrolizumab versus definitive RT followed by observation.

Exploratory Objectives:

Exploratory Objective #1:

* To determine the association of translational biomarkers including peripheral blood markers and tissue markers with patient outcomes.

Exploratory Objective #2:

* To determine changes in translational biomarkers including peripheral blood markers and tissue markers after receipt of definitive RT.

Exploratory Objective #3:

-To estimate PFS2, LRFS2, and DRFS2 in patients who crossed over from one randomization arm to the other arm.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for trial participation, patients must have:

1. The participant provides written informed consent for the trial.
2. Pathologically confirmed diagnosis of RCC with a clear cell component.
3. Be willing and able to undergo biopsy of a lesion planned for definitive RT. If a lesion amenable to SBRT was biopsied prior to enrollment, this material can be used in lieu of a planned biopsy if the tissue is available for review at MD Anderson.

   1. Patients may be allowed on this trial without a biopsy if they are deemed medically unfit for biopsy or if the biopsy poses undue risk in the opinion of the treating physician(s).
4. Be ≥18 years of age on the day of signing informed consent.
5. ECOG performance status 0-1.

NOTE: If subject is unable to walk due to paralysis, but is mobile in a wheelchair, subject is ambulatory for the purpose of assessing their performance status.

1. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
2. Oligometastatic RCC patients (≤5 metastatic lesions at the time of study entry). Per the discretion of the treating clinicians, we will not count lung lesions <1 cm short axis and LNs <1.5 cm short axis as these lesions are often equivocal.

   1. CNS disease will be allowed and the number of CNS lesions counted towards the number of metastatic lesions for the purposes of study entry.
3. Demonstrate adequate organ function as defined in the table below, all screening labs should be performed within 10 days prior to enrollment.
4. At least one site, which in the opinion of the treating radiation oncologist, is treatable with definitive RT and can be biopsied.
5. Criteria for known Hepatitis B and C positive subjects. Hepatitis B and C screening tests are not required unless:

   •Known history of HBV or HCV infection
   * As mandated by local health authority
6. Hepatitis B positive subjects • Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.

   • Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.
7. Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening.

   • Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization.

   Table Adequate Organ Function Laboratory Values System Laboratory Value --Hematological --Absolute neutrophil count (ANC) ≥1500/µL --Platelets ≥100 000/µL --Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La --Renal --Creatinine OR Measured or calculatedb creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN Hepatic --Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN --AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)

   --Coagulation International normalized ratio (INR) OR prothrombin time (PT)

   --Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

   --ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase);

   -- AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); ----GFR=glomerular filtration rate; ULN=upper limit of normal.

   a Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.

   b Creatinine clearance (CrCl) should be calculated per institutional standard. Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.

   Exclusion Criteria:

   The patient must be excluded from participating in the trial based on the following conditions:

1. The patient must have received their last dose of systemic therapy ≥24 weeks prior to initiation of their first dose of RT if this therapy included immunotherapy (e.g. pembrolizumab, nivolumab, ipilimumab, etc.) or ≥4 weeks prior to initiation of the first dose of radiation if this systemic therapy did not include immunotherapy.

2. Immunocompromising conditions, as follows:

* Known acute or chronic human immunodeficiency virus (HIV) infection
* History of primary immunodeficiency
* History of allogeneic tissue/solid organ transplant
* Current or prior use of immunosuppressive medication within 7 days before the first dose of study treatment, except for topical, ocular, intranasal, and inhaled corticosteroids, or systemic corticosteroids at an equivalent dose ≤10 mg of prednisone daily.

  3. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial as determined by the treating physician and/or member of the study team.

  4. Patients with a prior history of grade 3 or worse immune-related adverse events attributed to checkpoint inhibitors (PD-1, PD-L1, or CTLA-4), except endocrine adverse events with appropriate hormone replacement.

  5. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.

  6. Per the opinion of the treating physician of study team has cognitive impairments such that appropriate informed consent cannot be obtained or that he/she cannot participate in required study activities.
  1. Diffuse metastatic processes including leptomeningeal disease, diffuse bone marrow involvement, and peritoneal carcinomatous, which by the discretion of the treating physician cannot be treated definitively.
  2. Is pregnant, breast feeding, or expecting to conceive within the projected duration of the trial at the screening visit and at least one of the following conditions apply.
* Not a woman of childbearing potential (WOCBP) as defined in Appendix OR
* A WOCBP who agrees to follow the contraceptive guidance in Appendix during the treatment period and for at least 120 days (corresponding to time needed to eliminate any study treatment(s) (pembrolizumab and/or any active comparator/combination) plus 30 days (a menstruation cycle) after the last dose of study treatment.

  3. A WOCBP who has a positive urine pregnancy test within 72 hours prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Chad Tang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org